CLINICAL TRIAL: NCT07008716
Title: Omission of Clinical Target Volume (CTV) for Primary Tumors in Limited-Stage Small Cell Lung Cancer: A Prospective Multicenter Randomized Controlled Trial
Brief Title: Omitting CTV for Primary Tumor in LS-SCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shuohan Zheng, Dr., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-792
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: SCLC, Limited Stage; Radiation Exposure; Radiotherapy Side Effect; Progression
MeSH Terms: conditions — Radiation Injuries; Disease Progression | interventions — Radiotherapy; Etoposide; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Creating CTV for primary tumor.
  Interventions: Radiation: Radiation Therapy; Drug: Etoposide + carboplatin; Etoposide + cisplatin; Radiation: Creating CTV for primary tumor; Radiation: prophylactic cranial irradiation (PCI)
- Experimental group (Experimental): Omitting CTV for primary tumor.
  Interventions: Radiation: Radiation Therapy; Drug: Etoposide + carboplatin; Etoposide + cisplatin; Radiation: prophylactic cranial irradiation (PCI)

INTERVENTIONS:
Radiation: Radiation Therapy — Twice-daily (45 Gy/30 fractions) or once-daily (45 Gy/15 fractions) thoracic radiotherapy after 2-4 cycles of chemotherapy
Drug: Etoposide + carboplatin; Etoposide + cisplatin — Carboplatin IV (AUC=5) on day 1 combined with etoposide IV (100mg/m2) on days 1-3, or cisplatin IV (25mg/m2) on days 1-3 combined with etoposide IV (100mg/m2) on days 1-3. Treatment is repeated every 21 days for 4-6 cycles.
Radiation: Creating CTV for primary tumor — A margin of 0.8 cm beyond the gross target volume of primary tumor.
  Arms: Control group
Radiation: prophylactic cranial irradiation (PCI) — Beginning 4-6 weeks after chemoradiotherapy completion, patients in both arms who achieve a complete or partial response without brain metastasis receive PCI at 25 Gy/10 fractions or 26 Gy/13 fractions, delivered once daily (5 days per week).

SUMMARY:
This randomized controlled non-inferior trial prospectively enrolled patients with limited-stage small cell lung cancer (LS-SCLC). Patients in the experimental group would receive radiotherapy with omission of the clinical target volume (CTV) for the primary tumor, while those in the control group would receive radiotherapy including CTV. The efficacy and toxicity of the two groups are compared to provide evidence for the radiotherapy of LS-SCLC. The target volume of LS-SCLC may be reduced by omitting CTV without increasing local recurrence but potentially reducing the dose to organs at risk and the side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Small cell lung cancer confirmed by histology or cytology; TNM stage IA-IIIC (AJCC 8th edition, 2017; limited-stage) without intrapulmonary metastasis;
2. Aged 18-75 years, KPS score ≥ 80, ≤ 10% weight loss within the past 6 months;
3. Have measurable lesions per RECIST 1.1 criteria;
4. Have no disease progression after 2-4 cycles of etoposide/carboplatin or etoposide/cisplatin;
5. Lung function test: FEV1 ≥ 1 L (Optional);
6. Complete blood count: neutrophil count ≥ 1.5 x 10^9/L, hemoglobin ≥ 100 g/L, platelet count ≥ 100 x 10^9/L;
7. Renal function: serum creatinine ≤ 1.5 x upper limit of normal (ULN);
8. Liver function: AST and ALT ≤ 2.5 x ULN, bilirubin ≤ 1.5 x ULN;
9. Fully understand the study, able to complete treatment and follow-up, and voluntarily sign the informed consent.

Exclusion Criteria:

1. Other malignant tumors (prior or concurrent), except those that have been curatively treated with disease-free survival ≥ 5 years, such as non-melanoma skin cancer, cervical carcinoma in situ, or early-stage papillary thyroid cancer;
2. Uncontrolled heart disease or myocardial infarction within the past 6 months;
3. Patients with a history of mental illness;
4. Pregnant and lactating patients;
5. Poorly controlled diabetes and hypertension;
6. Interstitial pneumonia or active pulmonary fibrosis;
7. Active infection;
8. Other conditions unsuitable for enrollment (per investigator judgment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2025-06-03 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Local progression free survival | From the date chemotherapy commenced to the first clinical or radiological evidence of progressive disease at the primary site or death, whichever occurs first, to be assessed up to 3 years
Severe toxicity free survival | From the date chemotherapy commenced to the first record of serious adverse events related to radiotherapy, to be assessed up to 3 years

SECONDARY OUTCOMES:
Overall survival | From the date chemotherapy commenced to the date of death from any cause or the end of follow-up at 3 years
Progression free survival | From the date chemotherapy commenced to disease progression or death, whichever occurs first, to be assessed up to 3 years
Number of participants with recurrence or metastasis as evaluated by RECIST 1.1 | From the date chemotherapy commenced to the end of follow-up at 3 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the date chemotherapy commenced to the end of follow-up at 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhejiang Provincial Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No